CLINICAL TRIAL: NCT03355560
Title: A Single Arm Phase 2 Study of Adjuvant Nivolumab After Salvage Resection in Head and Neck Squamous Cell Carcinoma Patients Previously Treated With Definitive Therapy
Brief Title: Adjuvant Nivolumab After Salvage Resection in Head and Neck Cancer Patients Previously Treated With Definitive Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trisha Wise-Draper (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Trisha Wise-Draper, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-HN-17-01; CA209-997 (Other: Bristol Meyers Squibb)
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab starting 4-11 weeks after surgery for 6 doses.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 480 mg IV infusion
  Other Names: Opdivo

SUMMARY:
The purpose of this research study is to test the safety and efficacy of nivolumab after salvage resection in head and neck cancer in patients that have previously received definitive radiation with or without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Prior definitive therapy with radiation (with or without prior surgical resection and/or chemotherapy) who have underwent salvage resection with curative intent and have no other curable options
* Pre-operative scans including chest imaging preferably PET/CT and CT neck w/contrast. MRI neck is acceptable if contrast contraindicated.
* Able to provide archived biopsy or resected tissue.
* Adequate performance status and labs.

Exclusion Criteria:

* Patients who did not receive at least radiotherapy as prior definitive treatment.
* Patients who have gross measurable residual disease after surgery or those who underwent surgery for palliative purposes i.e. for symptom control.
* Has nasopharyngeal or sinonasal carcinoma.
* Has confirmed metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with Grade 3 and 4 adverse events of nivolumab | 28 weeks

SECONDARY OUTCOMES:
Percentage of patients any grade adverse events of nivolumab | 28 weeks
Disease free survival | 1 year
Disease free survival | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Wise-Draper, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - UC Health, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leddon JL, Gulati S, Haque S, Allen C, Palackdharry S, Mathews M, Kurtzweil N, Riaz MK, Takiar V, Nagasaka M, Patil Y, Zender C, Tang A, Cervenka B, McGrath J, Korn WM, Hinrichs BH, Jandarov R, Harun N, Sukari A, Wise-Draper TM. Phase II Trial of Adjuvant Nivolumab Following Salvage Resection in Patients with Recurrent Squamous Cell Carcinoma of the Head and Neck. Clin Cancer Res. 2022 Aug 15;28(16):3464-3472. doi: 10.1158/1078-0432.CCR-21-4554. PMID 35653116